CLINICAL TRIAL: NCT05119673
Title: Point-of-care Ultrasound for Difficult Peripheral Vascular Access in the Emergency Department - a Randomized Controlled Trial
Brief Title: POCUS for Difficult Peripheral Access in the Emergency Department - a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Butterfly Network (Industry)
Responsible Party: Principal Investigator, Emanuele Pivetta, Staff physician, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: POCUS-DiffAcc
Record Dates: First submitted 2021-10-20; First posted 2021-11-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Vascular Access; Emergencies
Keywords: Point-of-care ultrasound; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mono-plane sonographic view (No Intervention): Usual standard of care, in our institution, for difficult peripheral vascular access in the Emergency Department.
- bi-plane sonographic view (Active Comparator)
  Interventions: Other: bi-plane sonographic view to difficult peripheral vascular access using Butterfly iQ+®

INTERVENTIONS:
Other: bi-plane sonographic view to difficult peripheral vascular access using Butterfly iQ+® — Bi-plane Butterfly iQ+® sonographic visualization will be used to help Emergency Department operators to get a venous peripheral access in a population of patients considered difficult for this task based on their history or the present clinical situation.
  Arms: bi-plane sonographic view

SUMMARY:
Peripheral intravenous line insertion is the most commonly performed invasive procedure in the emergency department (ED). The research hypothesis is that a biplane sonographic approach (i.e., an out-of-plane and in-plane view) might be superior to a mono-plane approach (i.e., an out-of-plane or in-plane view) obtaining a peripheral vascular access among difficult patients admitted to the ED

DETAILED DESCRIPTION:
Peripheral intravenous line insertion is the most commonly performed invasive procedure in the emergency department (ED). In some studies, difficult vascular access population was about 33% of evaluated patients and for most of them the "blind" method (i.e., palpation) fails in the line insertion. Ultrasound guidance often increase the success rate among these patients.

Two basic techniques were proposed for sonographic guidance, a transversal or a longitudinal approach to the chosen vessel (i.e., out-of-plane or in-plane view, respectively, "mono-plane" approach).

The availability of hand-held sonographic devices is increasing the number of emergency department were this guidance is used in a difficult vascular access population.

The Butterly iQ+ device is now able to show out-of-plane and in-plane views, simultaneously, the so called bi-plane view.

Aim of this randomized controlled trial is to test if a bi-plane sonographic vision might be able to increase the performance of trained operators in obtaining a peripheral vascular access among difficult patients admitted to the ED.

The present study will be a randomized controlled, 2-arm, nonblinded trial held at the Città della Salute e della Scienza di Torino, University hospital, Turin, Italy.

All healthcare workers already trained in ultrasound-guided vascular access will be considered eligible for the study (i.e., emergency physicians, residents, nurses) after an ad hoc brief (2 hours) training on the study.

This will be a "real world" study, each provider will be free of choosing the device he/she thought appropriate for each patient (in terms of length, gauge, type - peripheral midline will be included in the Italian center).

Using a computerized permuted blocks of random sizes, enrolled patients will be randomized in a 1:1 ratio to be evaluated using either the "standard" ultrasound-guided approach (out-of-place or in-plane view) or the bi-plane view (i.e. out-of-place and in-plane view, simultaneously).

ELIGIBILITY:
Inclusion Criteria: at least one of the following criteria have to be present along with the need for a peripheral access

* chronic renal disease/ongoing dialysis;
* sickle cell anemia;
* prolonged and/or frequent use of i.v. drugs;
* difficult vascular access (after a first attempt or self-reported);
* previously need for more than one attempts / ultrasound guidance for getting a peripheral vascular access.

Exclusion Criteria:

* no consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
number of attempts of each peripheral i.v. access placement | Through study completion, likely of 1 year and half
  The number of attempts needed for getting a peripheral i.v. access will be measured
Time needed for each peripheral i.v. access placement | Through study completion, likely of 1 year and half
  Time needed for for getting a peripheral i.v. access will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Pivetta, MD,PhD, Principal Investigator — Città della Salute e della Scienza di Torino University Hospital
Locations (1):
- Emergency Department, Città della Salute e della Scienza di Torino Univeristy Hospital, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Result] Oliver WC Jr, Nuttall GA, Beynen FM, Raimundo HS, Abenstein JP, Arnold JJ. The incidence of artery puncture with central venous cannulation using a modified technique for detection and prevention of arterial cannulation. J Cardiothorac Vasc Anesth. 1997 Dec;11(7):851-5. doi: 10.1016/s1053-0770(97)90119-1. PMID 9412883
- [Result] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276
- [Result] Schummer W, Schummer C, Tuppatsch H, Fuchs J, Bloos F, Huttemann E. Ultrasound-guided central venous cannulation: is there a difference between Doppler and B-mode ultrasound? J Clin Anesth. 2006 May;18(3):167-72. doi: 10.1016/j.jclinane.2005.12.010. PMID 16731317
- [Result] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Comparison of three techniques for internal jugular vein cannulation in infants. Paediatr Anaesth. 2000;10(5):505-11. doi: 10.1046/j.1460-9592.2000.00554.x. PMID 11012954
- [Result] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Result] Keenan SP. Use of ultrasound to place central lines. J Crit Care. 2002 Jun;17(2):126-37. doi: 10.1053/jcrc.2002.34364. PMID 12096376
- [Result] Leung J, Duffy M, Finckh A. Real-time ultrasonographically-guided internal jugular vein catheterization in the emergency department increases success rates and reduces complications: a randomized, prospective study. Ann Emerg Med. 2006 Nov;48(5):540-7. doi: 10.1016/j.annemergmed.2006.01.011. Epub 2006 Feb 21. PMID 17052555
- [Result] Karakitsos D, Labropoulos N, De Groot E, Patrianakos AP, Kouraklis G, Poularas J, Samonis G, Tsoutsos DA, Konstadoulakis MM, Karabinis A. Real-time ultrasound-guided catheterisation of the internal jugular vein: a prospective comparison with the landmark technique in critical care patients. Crit Care. 2006;10(6):R162. doi: 10.1186/cc5101. PMID 17112371
- [Result] Augoustides JG, Horak J, Ochroch AE, Vernick WJ, Gambone AJ, Weiner J, Pinchasik D, Kowalchuk D, Savino JS, Jobes DR. A randomized controlled clinical trial of real-time needle-guided ultrasound for internal jugular venous cannulation in a large university anesthesia department. J Cardiothorac Vasc Anesth. 2005 Jun;19(3):310-5. doi: 10.1053/j.jvca.2005.03.007. PMID 16130056
- [Result] Troianos CA, Jobes DR, Ellison N. Ultrasound-guided cannulation of the internal jugular vein. A prospective, randomized study. Anesth Analg. 1991 Jun;72(6):823-6. doi: 10.1213/00000539-199106000-00020. No abstract available. PMID 2035868
- [Result] Mallory DL, McGee WT, Shawker TH, Brenner M, Bailey KR, Evans RG, Parker MM, Farmer JC, Parillo JE. Ultrasound guidance improves the success rate of internal jugular vein cannulation. A prospective, randomized trial. Chest. 1990 Jul;98(1):157-60. doi: 10.1378/chest.98.1.157. PMID 2193776
- [Result] Pittiruti M, Hamilton H, Biffi R, MacFie J, Pertkiewicz M; ESPEN. ESPEN Guidelines on Parenteral Nutrition: central venous catheters (access, care, diagnosis and therapy of complications). Clin Nutr. 2009 Aug;28(4):365-77. doi: 10.1016/j.clnu.2009.03.015. Epub 2009 May 21. PMID 19464090
- [Result] Troianos CA, Hartman GS, Glas KE, Skubas NJ, Eberhardt RT, Walker JD, Reeves ST; Councils on Intraoperative Echocardiography and Vascular Ultrasound of the American Society of Echocardiography. Guidelines for performing ultrasound guided vascular cannulation: recommendations of the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. J Am Soc Echocardiogr. 2011 Dec;24(12):1291-318. doi: 10.1016/j.echo.2011.09.021. No abstract available. PMID 22115322
- [Result] Maecken T, Grau T. Ultrasound imaging in vascular access. Crit Care Med. 2007 May;35(5 Suppl):S178-85. doi: 10.1097/01.CCM.0000260629.86351.A5. PMID 17446777
- [Result] Kumar A, Chuan A. Ultrasound guided vascular access: efficacy and safety. Best Pract Res Clin Anaesthesiol. 2009 Sep;23(3):299-311. doi: 10.1016/j.bpa.2009.02.006. PMID 19862889
- [Result] Chapman GA, Johnson D, Bodenham AR. Visualisation of needle position using ultrasonography. Anaesthesia. 2006 Feb;61(2):148-58. doi: 10.1111/j.1365-2044.2005.04475.x. PMID 16430568
- [Result] Ortega R, Song M, Hansen CJ, Barash P. Videos in clinical medicine. Ultrasound-guided internal jugular vein cannulation. N Engl J Med. 2010 Apr 22;362(16):e57. doi: 10.1056/NEJMvcm0810156. No abstract available. PMID 20410510
- [Result] French JL, Raine-Fenning NJ, Hardman JG, Bedforth NM. Pitfalls of ultrasound guided vascular access: the use of three/four-dimensional ultrasound. Anaesthesia. 2008 Aug;63(8):806-13. doi: 10.1111/j.1365-2044.2008.05513.x. Epub 2008 Jun 28. PMID 18549414
- [Result] Hopkins RE, Bradley M. In-vitro visualization of biopsy needles with ultrasound: a comparative study of standard and echogenic needles using an ultrasound phantom. Clin Radiol. 2001 Jun;56(6):499-502. doi: 10.1053/crad.2000.0707. PMID 11428801
- [Result] Venkatesan K. Echo-enhanced needles for short-axis ultrasound-guided vascular access. Int J Emerg Med. 2010 Apr 10;3(3):205. doi: 10.1007/s12245-010-0164-1. No abstract available. PMID 21031049
- [Result] Reynolds N, McCulloch AS, Pennington CR, MacFadyen RJ. Assessment of distal tip position of long-term central venous feeding catheters using transesophageal echocardiology. JPEN J Parenter Enteral Nutr. 2001 Jan-Feb;25(1):39-41. doi: 10.1177/014860710102500139. PMID 11190989
- [Result] Hsu JH, Wang CK, Chu KS, Cheng KI, Chuang HY, Jaw TS, Wu JR. Comparison of radiographic landmarks and the echocardiographic SVC/RA junction in the positioning of long-term central venous catheters. Acta Anaesthesiol Scand. 2006 Jul;50(6):731-5. doi: 10.1111/j.1399-6576.2006.01025.x. PMID 16987369
- [Result] Leyvi G, Taylor DG, Reith E, Wasnick JD. Utility of ultrasound-guided central venous cannulation in pediatric surgical patients: a clinical series. Paediatr Anaesth. 2005 Nov;15(11):953-8. doi: 10.1111/j.1460-9592.2005.01609.x. PMID 16238556
- [Result] Lamperti M, Caldiroli D, Cortellazzi P, Vailati D, Pedicelli A, Tosi F, Piastra M, Pietrini D. Safety and efficacy of ultrasound assistance during internal jugular vein cannulation in neurosurgical infants. Intensive Care Med. 2008 Nov;34(11):2100-5. doi: 10.1007/s00134-008-1210-9. Epub 2008 Jul 11. PMID 18618096
- [Result] Abboud PA, Kendall JL. Ultrasound guidance for vascular access. Emerg Med Clin North Am. 2004 Aug;22(3):749-73. doi: 10.1016/j.emc.2004.04.003. PMID 15301849
- [Result] Stone MB, Moon C, Sutijono D, Blaivas M. Needle tip visualization during ultrasound-guided vascular access: short-axis vs long-axis approach. Am J Emerg Med. 2010 Mar;28(3):343-7. doi: 10.1016/j.ajem.2008.11.022. Epub 2010 Jan 28. PMID 20223394
- [Result] Nichols I, Humphrey JP. The efficacy of upper arm placement of peripherally inserted central catheters using bedside ultrasound and microintroducer technique. J Infus Nurs. 2008 May-Jun;31(3):165-76. doi: 10.1097/01.NAN.0000317703.66395.b8. PMID 18496061
- [Result] Calvert N, Hind D, McWilliams R, Davidson A, Beverley CA, Thomas SM. Ultrasound for central venous cannulation: economic evaluation of cost-effectiveness. Anaesthesia. 2004 Nov;59(11):1116-20. doi: 10.1111/j.1365-2044.2004.03906.x. PMID 15479322
- [Result] Convissar D, Bittner EA, Chang MG. Biplane Imaging Versus Standard Transverse Single-Plane Imaging for Ultrasound-Guided Peripheral Intravenous Access: A Prospective Controlled Crossover Trial. Crit Care Explor. 2021 Oct 8;3(10):e545. doi: 10.1097/CCE.0000000000000545. eCollection 2021 Oct. PMID 34651134